CLINICAL TRIAL: NCT03737136
Title: Comparison Between Rituximab + PLX + IVIG With and Without Bortezomib in the Treatment of Antibody Mediated Kidney Transplanted Rejection
Brief Title: Comparison Between Bortezomib and Rituximab Plus Plasmapheresis in AMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMBU11254/B
Record Dates: First submitted 2018-11-04; First posted 2018-11-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Antibody-mediated Rejection
Keywords: transplantation; plasmapheresis
MeSH Terms: interventions — Bortezomib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasmapheresis (No Intervention): 5 Sessions Plasmapheresis and 100 mg/kg Intra venous immunoglobulin at the end of each session and one dose 375mg/m2 rituximab at the end of last session
- Plasmapheresis plus Bortezomib (Active Comparator): Drug 5 Sessions Plasmapheresis and 100 mg/kg Intra venous immunoglobulin at the end of each session and one dose 375ml/m2 rituximab at the end of last session plus bortezomib Injections 1.3mg/m2 intravenously on days 1, 4, 8, and 11
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — one cycle of bortezomib (each cycle: 1.3mg/m2 intravenously on days 1, 4, 8, and 11)
  Other Names: Velcade
  Arms: Plasmapheresis plus Bortezomib

SUMMARY:
Chronic-active antibody-mediated rejection (cAMR) due to de novo or pre-formed donor specific antibody (DSA) is currently considered the main cause of long-term allograft losses.Based on the aim of reducing or eliminating DSA, some proposed different therapeutic regimens for cAMR treatment. All of these protocols were derived from previous experience using acute antibody-mediated rejection and desensitization protocols, and mainly consisted of steroids, plasma exchange (PE), IVIG and RTX in various modalities. More recently, bortezomib was also proposed.To evaluate the role of a therapeutic regimen with plasma exchange, intravenous immunoglobulins and rituximab with or without Bortezomib in chronic-active antibody-mediated rejection (cAMR) settings this study designed.

DETAILED DESCRIPTION:
20 kidney transplant recipients (KTRs) with a diagnosis of cAMR in a prospective randomized clinical trial will be recruited in two arms

: ten KTRs treated with plasmapheresis, intravenous immunoglobulins and rituximab (PE-IVIG-RTX group) vs 10 patients receiving the same therapy plus Bortezomib. Differences between transplanted kidney survival and functional outcomes 6 mo after diagnosis and histological features and donor-specific antibody (DSA) characteristics (MFI ) will be investigated between two arms.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with renal biopsy demonstrating ABMR in the absence of T-cell-mediated rejection

Exclusion Criteria:

* Mixed AMR and T cell rejection
* do not sign the consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
graft survival | at month 6 following diagnosis
  Glomerular Filtration Rate

SECONDARY OUTCOMES:
Renal functional tests | at month 6 following diagnosis
  Serum Cr
Changes in Grading of antibody mediated rejection regarding Banff criteria in pathology | at month 6 following diagnosis
  kidney biopsy
DSAs-MFI | at month 6 following diagnosis
  Serum Test

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Beheshti MU sbmu, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- SBMU, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No